CLINICAL TRIAL: NCT07093736
Title: A Randomized Waitlist-controlled Trial to Evaluate of the Effectiveness of Immediate Treatment Compared to Deferred Treatment With the Fisher Wallace Stimulator FW-200 Device in First Responders With Self-reported Anxiety
Brief Title: A Study Comparing Immediate Treatment to Deferred Treatment With the Fisher Wallace (FW) Stimulator FW-200 Device for the Treatment of Self-reported Anxiety in First Responders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher Wallace Laboratories (Industry)
Collaborators: Advarra (Industry); Florence Healthcare (Unknown)
Responsible Party: Principal Investigator, Lois James, Ph.D., Associate Professor, WSU College of Nursing, Fisher Wallace Laboratories
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00053233
Record Dates: First submitted 2025-07-12; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Anxiety
Keywords: self-reported anxiety; first responder
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study was a waitlist-controlled study where the subjects were randomly assigned to receive an intervention immediately or after a specified delay. The two-week delay was designed to measure the natural progression of anxiety symptoms over a short period without intervention and to establish a baseline for how rapidly symptoms may escalate or impair functioning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Immediate treatment with FW-200 device (Experimental)
  Interventions: Device: FW-200
- Deferred treatment with FW-200 (Other): FW-200 treatment was delayed for two-weeks to measure the natural progression of anxiety symptoms over a short period without intervention and to establish a baseline for how rapidly symptoms may escalate or impair functioning.
  Interventions: Device: FW-200

INTERVENTIONS:
Device: FW-200 — Non-invasive, home-use neurostimulation device delivering transcranial fixed output, alternating current stimulation

SUMMARY:
The goal of this clinical trial is to learn if the Fisher Wallace Stimulator FW-200 experimental device is effective at treating self-reported anxiety in first responders. The main question the trial aims to answer is does the FW-200 device improve anxiety as measured by a validated questionnaire.

DETAILED DESCRIPTION:
This is a randomized waitlist-controlled trial to evaluate the efficacy and safety of the Fisher Wallace Stimulator FW-200 device in the treatment of self-reported anxiety in police personnel and first responders. Participants will be randomly assigned to receive immediate treatment or deferred treatment with the FW-200 device.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Ability to read and write in English
* First responder employee or employee of participating police department
* Beck Anxiety Inventory total score above 7
* Able to commit to two 20-minute device treatment session per day for up to 8 weeks
* Willing to wear an actigraphy device

Exclusion Criteria:

* Use of brain stimulation device in the last year
* Have a pacemaker, electronic stent or electronic implants
* Started or planning to start new medial treatment or health program over the next 8 weeks
* Contemplated suicide in the past year
* Institutionalized for mental health issues
* Have a serious medical condition
* Currently taking medications affecting the nervous system
* Allergic to nickel
* Currently taking or planning to take part in any other study on insomnia, anxiety or other mental health effort over the next 8 weeks
* Currently pregnant or planning to become pregnant in the next 10 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory (BAI) scores | From baseline to week 2
  Change in Beck Anxiety Inventory (BAI) scores at Week 2 versus baseline in immediate treatment group compared to the deferred treatment group. Total score range is a minimum of 0 to a maximum of 63. Higher score means a worse severity of anxiety.

SECONDARY OUTCOMES:
Patient Health Questionnaire | From baseline to week 2 and week 4. Total scores range from 0 to 24. Higher scores mean worse severity of depressive symptoms.
  Change in Patient Health Questionnaire-8
Professional Quality of Life | From baseline to week 2 and week 4
  Change in Professional Quality of Life
Consenting to Study Continuation | Week 4
  Percentage of participants consenting to study continuation at week 4 in the immediate treatment group compared to deferred treatment group
Total Sleep Time | Baseline to through study completion
  Percentage of participants with a 20 minute or more increase in total sleep time for the immediate treatment group compared to the deferred treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Lois James, Ph.D., Principal Investigator — James Consulting
Locations (2):
- United States (2):
  - Florence Healthcare, Atlanta, Georgia
  - Seattle Police Department Wellness Unit, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided